CLINICAL TRIAL: NCT05248711
Title: Testing the Feasibility of Brief Daily App-Based Mindful Movements in US Adults
Brief Title: Project Movement/Daily Move Feasibility
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Personnel Change
Sponsor: Calm.com, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Calm2021-105
Record Dates: First submitted 2022-01-19; First posted 2022-02-21 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Stress

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily Move (Experimental): Participants (n=107) will be provided free access to and asked to register for the consumer-based mobile meditation app, Calm, on their phone. Participants will then receive an email containing one year of free access to Calm. Participants will be asked to use the Daily Move component on the Calm app for ~10 minutes per day for 8 weeks.
  Interventions: Behavioral: Calm Daily Move
- Usual Care (No Intervention): Participants (n=107) will be asked to continue with usual care/routine and complete survey measures at each time point. Participants will be provided with access to the intervention after their study participation.

INTERVENTIONS:
Behavioral: Calm Daily Move — The Daily Move is a series of short, 5-min videos outlining mindful movement exercises. The Daily Move is part of the Calm app's library of content.
  Arms: Daily Move

SUMMARY:
The purpose of this study is to test the feasibility (acceptability and demand) of the Daily Move in a diverse sample of US adults. Acceptability benchmarks: 214 participants recruited within three months (60% will identify as a racial/ethnic minority; 30% African American, 30% Hispanic); At least 70% of participants rate the intervention as satisfactory. Demand benchmarks: At least 70% of participants complete 75% of prescribed Daily Move sessions per week across the 8-weeks; Dropouts not to exceed >30% of participants. Aim 2 - explore the pre-post trends in change of: Stress - Perceived Stress Scale (PSS), Anxiety and Depression - Hospital Anxiety and Depression Scale (HADS), Mindfulness- Mindful Attention Awareness Scale (MAAS), and Mood- Profile of Mood States (POMS).

DETAILED DESCRIPTION:
Generalized stress among adults is an increasingly problematic concern, particularly in recent years due to the COVID-19 pandemic. According to the Stress in America 2020 data, Americans are still struggling to cope with the disruptions that the pandemic has caused, and nearly 8 in 10 adults (78%) say that the COVID-19 pandemic is a significant source of stress in their life. This stress from the COVID-19 pandemic is in addition to previous sources of stress that impacted American adults, including things such as health care, mass shootings, global climate change, and more. Additionally, rising concerns over racism and racially-driven acts of violence has impacted racial-ethnic minorities and led to rising rates of stress over discrimination. In 2021, 44% of people of color said that discrimination was a significant source of stress in their life, compared with 38% back in 2019. The currently proposed study aims to include American adults with elevated levels of stress, with 60% of the recruited sample targeting racial-ethnic minorities.

The investigators have previously conducted multiple feasibility and pilot studies investigating the use of the mobile meditation app, Calm, on various mental health outcomes in a diverse range of adults (cancer patients, adults with sleep disturbances, etc.). The investigators have found the Calm meditation app to be both feasible and beneficial for adults on a range of mental health outcomes, including stress-related outcomes. Although there is a growing body of evidence to describe the benefits of short, daily meditations on stress and other mental health outcomes in adults, there are currently no investigations that have been done to examine the feasibility or impact of short, daily app-based mindful movement exercises on stress in adults. It is for these reasons that the primary purpose of this study is to test the feasibility of the Calm's "Daily Move" component on stressed adults.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Score of 6 or greater on the Perceived Stress Scale-4

Exclusion Criteria:

* Subscribe to Calm or use Calm
* Live outside of the United States of America
* Unable to read or understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Stress | Changes in stress will be measured at baseline, week 2, week 4, week 6, and week 8 (post-intervention). The PSS includes 10 items with total scores ranging from 0-40.
  Stress will be measured using the Perceived Stress Scale (PSS).

SECONDARY OUTCOMES:
Anxiety | Changes in anxiety will be measured at baseline, week 4, and week 8 (post-intervention). The HADS includes seven items assessing anxiety symptoms with a total score range of 0-21.
  Anxiety will be measured using the Hospital Anxiety and Depression Scale (HADS).
Depression | Changes in depression will be measured at baseline, week 4, and week 8 (post-intervention). The HADS includes seven items assessing depressive symptoms with a total score range of 0-21.
  Depression will be measured using the Hospital Anxiety and Depression Scale (HADS).
Mindfulness | Changes in mindfulness will be measured at baseline, week 4, and week 8 (post-intervention). The MAAS is a 15-item scale with total possible scores ranging from 15-90, with higher scores indicating greater mindfulness.
  Mindfulness will be measured using the Mindful Attention Awareness Scale (MAAS).
Mood | Changes in mood will be measured at baseline, week 4, and week 8 (post-intervention). The POMS is a 65-item scale with six sub scales. Each item is scored on a 0-4 scale, yielding a total possible score range of -24 to 177.
  Mood will be measured using the Profile of Mood States (POMS).

OTHER OUTCOMES:
Study Satisfaction | Study satisfaction will be measured at week 8 (post-intervention).
  Study satisfaction will be measured using an investigator-developed satisfaction survey.

CONTACTS AND LOCATIONS:
Overall Officials: Calm, Study Director — Calm.com, Inc.
Locations (1):
- Calm, Inc., San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No